CLINICAL TRIAL: NCT03299829
Title: A Retrospective Study to Assess the Clinical Efficacy and Safety of Trientine in Wilson's Disease Patients
Status: Completed | Type: Observational
Sponsor: Excelsior (Industry)
Responsible Party: Sponsor
Other Study IDs: EB-TR-001
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Trientine Treatment for Wilson's Disease
Keywords: trientine; Wilson's disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Trientine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Trientine — Trientine is a chelating agent for removing the copper from the body

SUMMARY:
This is a retrospective study to assess the clinical efficacy and safety of trientine in Wilson's disease patients

DETAILED DESCRIPTION:
In this retrospective study, the investigators will collect and analyze data from reviewing medical history files of larger and long-term follow-up cohorts with Wilson's disease in Taiwan to assess the efficacy and safety of Trientine in Taiwanese Wilson's Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Wilson's disease.
* Male or female patients, aged 3 years to 75 years

Exclusion Criteria:

* Patients with comorbidity which is not related to Wilson's disease.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had the diagnosis of Wilson's disease
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The improvement in liver function | Up to 1 year
  To measure the AST (aspartate aminotransferase), ALT (alanine transaminase), GGT (gamma-glutamyl transpeptidase), Albumin, and Bilirubin level, and compare to the baseline

SECONDARY OUTCOMES:
The improvement in urine copper excretion | Up to 1 year
  To measure 24-hour urine copper levels during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Chinchang Huange, Doctor, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Linkou, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No